CLINICAL TRIAL: NCT04435912
Title: The Role of Hydrocortisone Per-treatment in Decreasing Side Effects of Protamine Sulfate During Cardiac Surgeries, a Randomized Control Trial.
Brief Title: Hydrocortisone Per-treatment Decrease Side Effects of Protamine Sulfate
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Mustafa Alrabayah, Assistant Professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MAlrabayah
Record Dates: First submitted 2020-06-09; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Blood Pressure; Heart Rate; Airway Pressure
Keywords: Protamine sulfate; Hydrocortisone; Protamine Sulfate side effects
MeSH Terms: interventions — Hydrocortisone

STUDY DESIGN:
Intervention Model Description: Parallel group, randomized, controlled trial with 1:1 allocation ratio. Participants were Patients undergoing cardiac surgery using cardiopulmonary bypass.
Who Masked: Care Provider, Investigator
Masking Description: Randomization envelopes kept closed until the completion of patient registration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PS alone group (No Intervention): Patients received only Protamine Sulfate for reversal of Heparin
- PS and HC group (Experimental): Patients received Hydrocortisone pre-treatment then Protamine Sulfate for the reversal of Heparine
  Interventions: Drug: Hydrocortisone 200mg IV

INTERVENTIONS:
Drug: Hydrocortisone 200mg IV — single dose pre-treatment given IV given at the time when the patient is attached to the cardiopulmonary bypass machine
  Arms: PS and HC group

SUMMARY:
This study aims to compare the hemodynamic parameters within and between patients who received Protamine Sulfate (PS) with Hydrocortisone (HC) vs. Protamine Sulfate alone during cardiac surgeries.

DETAILED DESCRIPTION:
the investigators hypothesized that patients received PS along with HC would have different results in intraoperative hemodynamic changes of the blood pressure - both Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP) and Mean Arterial Pressure (MAP) reading. Differences would also be expected for Heart rate (HR), Airway pressure and the usage of Adrenaline, Noradrenaline and Dobutamine.

Patients who had cardiac surgery using cardiopulmonary bypass were screened and enrolled from 4/7/2019 to 30/4/2020. Inclusion criteria for patients were normal preoperative hemoglobin level, normal preoperative platelet count, no known defect of the coagulation system, and patients with unimpaired renal function (creatinine clearance < 30 ml/kg/min). The patients were excluded if they were younger than 18 years, patients with known defect of the coagulation system, renal impairment, previous vasectomy, allergy to fish or unable to give consent form.

The study carried out as a parallel-group, randomized, controlled trial with a 1:1 allocation ratio. Patients were screened for eligibility in the wards before being invited to participate in the research. After the invitation, the study was explained to patients. Those who agreed to participate in the study were asked to sign the consent form.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had cardiac surgery using cardiopulmonary bypass
* Normal preoperative hemoglobin level
* Normal preoperative platelet count
* No known defect of the coagulation system
* Patients with unimpaired renal function (creatinine clearance < 30 ml/kg/min)

Exclusion Criteria:

* Patients younger than 18 years
* Patients with known defect of the coagulation system
* Renal impairment
* Previous vasectomy
* Allergy to fish
* Unable to give consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure | changes of baseline blood pressure taken preoperatively and readings taken during 30 minutes after Protamine Sulfate was given
  both systolic, diastolic and mean arterial pressure

SECONDARY OUTCOMES:
Hemodynamic parameters | changes of baseline readings taken preoperatively and readings taken during 30 minutes after Protamine Sulfate was given
  Heart rate (Beat Per Minute),
Hemodynamic parameters | changes of baseline readings taken preoperatively and readings taken during 30 minutes after Protamine Sulfate was given
  Airway pressure (cm H2O)
Hemodynamic parameters | the change in drugs doses required to maintain mean arterial pressure more than 65 mmHg during the first 30 minutes following Protamine dose
  The usage of Adrenaline, Noradrenaline and Dobutamine (microgram/kg/min).

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa A Alrabayah, MD, Study Director — The University of Jordan
Locations (1):
- Faculty of Medicine, Zarqa, Jordan

IPD SHARING:
Plan to Share IPD: No
decision depends on the roles and regulations of The University of Jordan